CLINICAL TRIAL: NCT06493591
Title: Atrial Fibrillation Ablation and Autonomic Modulation Via Thoracoscopic Surgery, 10 Year Follow up.
Acronym: AFACT-10
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, J.R. de Groot, Principal Investigator, Professor of electrophysiology, Amsterdam UMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL87358.018.24
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Thoracoscopy; Ganglia, autonomic; Ganglion Plexus; Ablation
MeSH Terms: conditions — Atrial Fibrillation; Ganglion Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subgroup: GP ablation: Participants underwent thoracoscopic AF ablation with additional GP ablation as the intervention group in the AFACT study.
  PVI with additional left atrial ablation lines was performed and conduction block was verified.
  No additional intervention will be perforemd in this study. All study procedures will be the same for the two subgroups.
- Subgroup: No GP ablation: Participants underwent thoracoscopic AF ablation as the control group in the AFACT study.
  PVI with additional left atrial ablation lines was performed and conduction block was verified.
  No additional intervention will be perforemd in this study. All study procedures will be the same for the two subgroups.

SUMMARY:
This observational study investigates the long-term outcomes of patients ten years after their participation in a previous study on the surgical treatment of atrial fibrillation (AF). Participants were part of a the AFACT study a decade ago that explored whether damaging nerves around the heart could reduce AF. Participants were randomized to standard thoracoscopic AF ablation (MiniMaze) with or without Ganglion Plexus (GP) ablation. This new study aims to assess and compare the long-term effects of these treatments. We are specifically interested which treatment leads to more freedom from AF.

Key questions include:

How many patients are free from AF ten years after treatment without using antiarrhythmic drugs? What are the complications from both treatments?

Participants will undergo the following assessments:

* Clinical assessment at the outpatient clinic.
* ECG and 24-hour Holter ECG
* Echocarddiogram and laboratory assessment.
* SF-36 Quality of life questionnaire.

DETAILED DESCRIPTION:
Rationale: Invasive treatment of atrial fibrillation (AF) has a limited efficacy. A substantial group of patients keep having symptoms of AF after ablation. Autonomic modulation of AF through ablation of the ganglion plexi (GP) has been suggested as an addition to surgical AF ablation. The AFACT trial demonstrated futility of GP ablation added to thoracoscopic ablation of AF at 1 and 2 years follow-up. Long term efficacy and safety of autonomic modulation of AF is unknown.

Objective: To evaluate the efficacy and safety of GP ablation in addition to thoracoscopic PVI after 10 years of follow-up in patients with advanced AF.

Study design: This single center cohort study will re-investigate participants in the AFACT trial. The study consists of three parts. First, a national mortality database examination will be conducted to identify the participants in AFACT who died in the last 10 years. Second, a prospective clinical assessment at the outpatient clinic and third a retrospective chart review. Patients will be invited to a single visit at the outpatient clinic to sign informed consent and a subsequent clinical assessment by an investigator. Additionally, patients will be examined through a 12-lead electrocardiogram(ECG), a 24-hour holter ECG, transthoracic echo (TTE), laboratory assessment and they will be asked to complete the SF-36 quality of life (QOL) questionnaire. Furthermore, a retrospective chart review will be performed integrating data from the AFACT trial with subsequent clinical information obtained through medical chart reviews were we will focus on finding the first recurrence of AF.

Study population: The study population comprises participants from the AFACT trial, who were adults who underwent thoracoscopic ablation for advanced atrial fibrillation (AF). In the AFACT trial 240 patients were randomized to thoracoscopic ablation + GP ablation or thoracoscopic ablation.

Intervention (if applicable): N.A. Main study parameters/endpoints: 1: Freedom of AF ten years after the procedure without the use of antiarrhythmic drugs. 2: Time to first AF recurrence. 3: Type of AF recurrence, i.e. paroxysmal, persistent and permanent AF and atrial tachycardia (AT). 4: Left atrial (LA) volume and function. 5: QOL. 6: Pacemaker implants. 7: Additional ablation procedures. 8: Major adverse events.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The benefit of this study is that patients have an extra control visit to investigate the heart rhythm and that physical examination is performed, if necessary. This study carries no risks for the patients.

ELIGIBILITY:
Inclusion Criteria:

* AFACT Trial participant

Exclusion Criteria:

* Refusal to be contacted for future studies during or since the AFACT trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises participants from the AFACT trial, all of whom underwent thoracoscopic ablation for advanced AF. The AFACT trial encompassed 240 patients that underwent thoracosopic AF ablation for persistent AF, enlarged left atria (left atrial volume index [LAVI] >33 ml/m2), prior unsuccessful catheter ablation, or patient preference for thoracoscopic ablation. Patients had a mean age at time of inclusion of 59.9 +-8.2 years and 73% of participants were male. Importantly, the surgical ablation occurred approximately 10 years ago for for all participants. During the AFACT trial, 4 out of the 240 patients died, leaving a maximum of 236 patients for this analysis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Freedom of AF | 10 years
  Number of participants with freedom of AF after ten years after the procedure without the use of antiarrhythmic drugs. Freedom of AF is defined as the absence of documentation of episodes of AF, atrial flutter or atrial tachycardia >30 seconds on all holters and ECG recordings during follow up.

SECONDARY OUTCOMES:
Time to first AF recurrence. | Within 10 year follow up.
  Time to first AF recurrence defined as the first documentation of documentation of AF >30 seconds during follow up.
Classification of AF recurrence | 10 years
  Classifications of AF recurrence and change from baseline of AF recurrence classification (paroxysmal, persistent, permanent AF, and atrial tachycardia).
Left Atrial Volume and Function | Between 8 and 10 years follow up
  left Atrial (LA) Volume and Function 8 to 10 years post procedure compared between the two arms. And the change in Left Atrial (LA) Volume and Function from baseline to 8 to 10 years post procedure compared.
Quality of Life improvement | 10 years
  Improvement from baseline of functional status as measured by the RAND 36 quality of life questionnaires at 10 years
Pacemaker implants | 10 years
  Number and reasons for pacemaker implants during the ten-year follow-up period.
Additional ablation | 10 years
  Number and reasons for additional ablation procedures during the ten-year follow-up period.
Cardioversions | 10 years
  Number and reasons for cardioversions during the ten-year follow up.
Major cardiovascular adverse events | 10 years
  Occurrence of major adverse events (heart failure, stroke, major bleeding, mortality) during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. J.R. de Groot, Principal Investigator — Amsterdam UMC